CLINICAL TRIAL: NCT03161886
Title: A Treat-to-target Strategy Using Pan-enterica Capsule Endoscopy (PCE) in Paediatric Crohn's Disease (CD).
Brief Title: A Treat-to-target Strategy Using Pan-enteric Capsule Endoscopy (PCE) in Paediatric Crohn's Disease (CD).
Acronym: PCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Salvatore Oliva, Research Assistant, Azienda Policlinico Umberto I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCE Monitoring CD
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Bowel Diseases; Children, Only
Keywords: colon capsule endoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pan-enteric capsule endoscopy (PCE) (Experimental): Evidence of active disease by PCE prompted a change in therapy at the discretion of the treating clinician and according to current available pediatric guidelines. The definition of medical treatment adjustment after evidence of inflammation was: the introduction of steroids or enteral nutrition, the introduction or optimization of immunosuppressives; the introduction, optimization of biologics; or the introduction of both immunosuppressive agents and biologics. In case of a negative PCE and presence of symptoms, the magnetic resonance enterography (MRE) could help in guiding therapeutic decisions.
  Interventions: Device: Pan-enteric Capsule Endoscopy (PCE)

INTERVENTIONS:
Device: Pan-enteric Capsule Endoscopy (PCE) — Second generation of colon capsule endoscopy (Medtronic)

SUMMARY:
This prospective, interventional study aims this to determine the efficacy and safety of a PCE-based treat-to-target strategy in order to achieve Mucosal Healing (MH) and deep remission (DR) of pediatric Crohn's Disease (CD) over 52 weeks.

DETAILED DESCRIPTION:
This first prospective study on mucosal healing (MH) and deep remission (DR) in pediatric Crohn's Disease aims to evaluate:

* The ability of Pan-enteric capsule endoscopy (PCE) to assess MH and DR rates at three time points and to guide a treat-to-target strategy was the primary outcome sought.
* The efficacy of a "treat-to-target" strategy to MH and DR rates over 24 and 52 weeks was evaluated as a secondary outcome;
* Comparison between PCE, biomarkers, Magnetic Resonance Enterography (MRE) and Small Intestine contrast ultrasonography (SICUS) in evaluating intestinal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Crohn's Disease made at least 3 months before the enrolment;
* subject was referred for endoscopic and imaging follow-up in Crohn's Disease
* signed informed consent.

Exclusion Criteria:

* Subject has dysphagia
* Subject has renal insufficiency
* Subject is known structuring Crohn's Disease identified by magnetic resonance enterography (MRE) or small intestine contrast ultrasonography (SICUS).
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the magnetic resonance enterography findings and clinical judgment of the investigator.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Monitoring mucosal healing | 52 weeks
  -The ability of PCE to assess mucosal healing rate (percentage of patients with healing of the mucosa) at three time points and to guide a treat-to-target strategy was the primary outcome sought.
  and colonic CD
Monitoring deep remission | 52 weeks
  -The ability of PCE to assess deep remission rate (percentage of patients with healing of the mucosa and absence of symptoms) at three time points and to guide a treat-to-target strategy was the primary outcome sought.
  and colonic CD

SECONDARY OUTCOMES:
Treat to Target | 52 weeks
  -The efficacy of a "treat-to-target" strategy to increase percentage of patients with mucosal healing (healing of the mucosa) and deep remission (healing of the mucosa and absence of symptoms) rates over 24 and 52 weeks
Diagnostic Yield | 52 weeks
  percentage of patients with positive finding at PCE, biomarkers, Magnetic Resonance Enterography (MRE) and Small Intestine contrast ultrasonography (SICUS).

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Oliva, MD, Principal Investigator — Sapienza - University of Rome, Azienda Policlinico Umberto I

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oliva S, Cucchiara S, Civitelli F, Casciani E, Di Nardo G, Hassan C, Papoff P, Cohen SA. Colon capsule endoscopy compared with other modalities in the evaluation of pediatric Crohn's disease of the small bowel and colon. Gastrointest Endosc. 2016 May;83(5):975-83. doi: 10.1016/j.gie.2015.08.070. Epub 2015 Sep 9. PMID 26363334
- [Derived] D'Arcangelo G, Russo G, Aloi M, Ruggiero C, Maccioni F, Hassan C, Papoff P, Cohen SA, Oliva S. A Treat-to-Target Strategy Guided by Pan-Enteric Evaluation in Children With Crohn's Disease Improves Outcomes at 2 Years. Inflamm Bowel Dis. 2024 Aug 1;30(8):1303-1308. doi: 10.1093/ibd/izad173. PMID 37603835
- [Derived] Oliva S, Aloi M, Viola F, Mallardo S, Civitelli F, Maccioni F, Hassan C, Papoff P, Cucchiara S, Cohen SA. A Treat to Target Strategy Using Panenteric Capsule Endoscopy in Pediatric Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2060-2067.e1. doi: 10.1016/j.cgh.2018.10.015. Epub 2018 Oct 13. PMID 30326301